CLINICAL TRIAL: NCT01025492
Title: Mechanisms of Atheroprotection by Fenofibric Acid (ABT 335) Added to a Statin in Subjects With Insulin Resistance (Hypertriglyceridemia and Low HDL-C)
Brief Title: Study of Trilipix Effects on Lipids and Arteries
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Collaborator/corporate sponsor withdrew funding and permission to continue.
Sponsor: University of Utah (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00030151
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-07

CONDITIONS: Dyslipidemia
Keywords: high density lipoprotein; arterial compliance; brachial artery flow-mediated dilatation
MeSH Terms: conditions — Dyslipidemias | interventions — Fenofibrate; fenofibric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trilipix (Active Comparator): Trilipix (fenofibric acid) 135 mg tablet orally, once daily for 12 weeks
  Interventions: Drug: Trilipix
- Placebo (Placebo Comparator): Matching placebo tablet orally, once daily for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Trilipix — 135 mg po daily
  Other Names: fenofibric acid
  Arms: Trilipix
Drug: placebo — one tablet po daily
  Arms: Placebo

SUMMARY:
Fibrates reduce atherosclerosis and cardiovascular disease events. A major mechanism of this benefit appears to be their ability to raise plasma high density lipoprotein cholesterol (HDL-C), especially in patients with high triglyceride levels. This study will investigate the effects of the addition of Trilipix (fenofibric acid) versus placebo to ongoing statin treatment on high density lipoprotein (HDL) composition and arterial function in subjects with insulin resistance.

DETAILED DESCRIPTION:
The field of lipid treatment for atheroprevention, and of HDL-raising in particular, was shaken by the unexpected finding of a net adverse clinical effect of torcetrapib, a Cholesteryl ester transfer protein (CETP) inhibitor with HDL-raising effects far more dramatic than that of niacin or fenofibrate.

Trilipix (ABT 335, choline fenofibrate, or fenofibric acid) is approved by the FDA (12/2008) for treatment of dyslipidemia and may act as a new fibrate for treatment of dyslipidemia and atheroprevention. It is the first fibrate with sufficient evidence for safety in combination use with a statin to receive an FDA indication for that combination use. Thus, there is minimal safety risk to prospective research subjects, who in any case will have the very dyslipidemia for which this combination is approved and recommended. With the ongoing development of this agent through a time of great scientific controversy regarding torcetrapib and HDL, it is urgent to explore the HDL-related mechanisms by which Trilipix may be atheroprotective, with special attention to changes in HDL composition and function.

Novel methods have been developed for measuring HDL composition and function and have been added to state-of-the-art technologies to assemble the uniquely comprehensive panel of HDL parameters in this study. Such methods can now be employed in exploring potentially beneficial effects of promising HDL-active agents such as Trilipix. In addition, improvements in HDL with fibrates appear to be related to other favorable lipoprotein changes, such as reduced remnant levels and increased LDL particle size, and these likely help explain arterial benefits with these agents.

The recent advent and validation of many non-invasive methods for measuring arterial function allows characterization of arterial effects of lipid agents in a time- and cost-effective way, alternative to standard event-driven trials. This study offers a uniquely comprehensive panel of these arterial parameters in order to characterize the likely atheropreventive effects of Trilipix.

This study will investigate changes in both panels of endpoints (state-of-the-art measures of HDL and related lipoproteins, and of arterial function) with Trilipix, which will more clearly and broadly define the benefits of this agent than has been done for any other lipid therapy. In addition, analyses of the intercorrelations of the changes among these several parameters should strongly suggest mechanisms of atheropreventive benefits of Trilipix.

Finally, with regard to subject selection, most patients with insulin resistance are at high risk for atherosclerosis, even those without concurrent diabetes mellitus. Importantly, favorable effects of fibrates are most pronounced in patients with insulin resistance, whether manifested traditionally by central obesity, adiposity, glucose and insulin abnormalities. Beta-cell dysfunction, generally seen in conjunction with insulin resistance, might also predict benefit with fibrate therapy. Body composition (as adiposity or central obesity) is a strong correlate of these abnormalities and will be measured during the study. Already at present, and more so in the future, the standard of care for insulin resistant patients will be statin monotherapy. In addition, however, fibrates are being increasingly advocated as adjunctive therapy for patients with residual abnormalities of triglyceride and HDL-C after statin monotherapy. Thus, the best way to assess the likely benefits of Trilipix in the usual clinical practice setting is to do so against a background of stable statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Triglyceride 150-500 mg/dL
* HDL-C < 45 mg/dL in men, < 55 in women
* LDL-C < 130 mg/dL
* stable statin dose x 8 weeks

Exclusion Criteria:

* Prior use of a fibrate > 4 weeks ever (minimum 12 months off fibrate)
* Intolerance to medications to be used in study (fenofibric acid, albuterol, nitroglycerin)
* Niacin or thiazolidinedione within the prior 12 months, or anticipated need to add either during 6-month study period
* Diabetes Mellitus if either (1) diagnosed less than 3 months ago, (2) treated with insulin, or (3) with an A1c >8%
* Anticipated need to change treatment regimen of statin (or other lipid agent) or glycemic treatment during 6-month study period
* Uncontrolled hypertension (BP > 140/90 mm Hg), or changes in BP meds within prior 4 weeks, or anticipated need to change BP meds during 6-month study period
* Documented cardiovascular disease event (heart attack, stroke, or hospitalization for unstable angina or revascularization procedure) in the past 6 months
* Use of warfarin (potential to interact adversely with fibrate therapy)
* Uncontrolled thyroid disease (TSH outside of normal range)
* Renal insufficiency (calculated Glomerular Filtration Rate <50 ml/min)
* Hepatic disease (ALT > 1.5x Upper Limit of Normal, diagnosis of hepatitis, cirrhosis)
* Active cholecystitis/cholelithiasis
* Active cancer (except basal cell or squamous cell skin cancer)
* Pregnancy, plan/desire to become pregnant, breast feeding
* Inability or unwillingness to provide informed consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliot Brinton, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The clinical trial collaborator/corporate sponsor prematurely terminated the study and did not provide unblinding information to the investigator or study team, therefore it is not known to which arm/group each of the participants enrolled.
Groups:
- Trilipix or Placebo: Trilipix - 135 mg tablet orally, once daily for 12 weeks; or Placebo - matching placebo tablet orally, once daily for 12 weeks
Period: Overall Study
Arm/Group | Trilipix or Placebo
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The clinical trial collaborator/corporate sponsor prematurely terminated the study and did not provide unblinding information to the investigator or study team. It is not known to which arm/group each of the participants enrolled, therefore all enrolled subjects were included in a single arm/group.
Arm/Group | Trilipix or Placebo
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Apolipoprotein A-I Serum Concentration
Description: Comparison of apolipoprotein A-I concentrations after 12 weeks of treatment with either Trilipix or placebo
Time Frame: 12 weeks
Population: The clinical trial collaborator/corporate sponsor prematurely terminated the study and did not provide unblinding information to the investigator or study team, therefore it is not known to which arm/group each of the participants enrolled. Additionally, the study outcome measure/endpoint (Apolipoprotein A-I serum concentration) was not analyzed.
Arm/Group | Trilipix or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: The clinical trial collaborator/corporate sponsor prematurely terminated the study and did not provide unblinding information to the investigator or study team, therefore it is not known to which arm/group each of the participants enrolled.
Arm/Group | Trilipix or Placebo
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No